CLINICAL TRIAL: NCT02700230
Title: Phase I Trial of Intratumoral Administration of a NIS-Expressing Derivative Manufactured from a Genetically Engineered Strain of Measles Virus in Patients with Unresectable or Recurrent Malignant Peripheral Nerve Sheath Tumor
Brief Title: Vaccine Therapy in Treating Patients with Malignant Peripheral Nerve Sheath Tumor That is Recurrent or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1372; NCI-2016-00179 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1372 (Other: Mayo Clinic); W81XWH-15-1-0115 (Other Grant/Funding Number: Department of Defense); 15-008308 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-02-25; First posted 2016-03-07 (Estimated); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Malignant Peripheral Nerve Sheath Tumor; Neurofibromatosis Type 1; Recurrent Malignant Peripheral Nerve Sheath Tumor
MeSH Terms: conditions — Neurofibrosarcoma; Neurofibromatosis 1 | interventions — X-Rays; Photons; Magnetic Resonance Spectroscopy; High-Energy Shock Waves; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (MV-NIS) (Experimental): Patients receive MV-NIS intratumorally on day 1. Patients also undergo SPECT/CT at baseline and at 3 and 8 days after MV-NIS. Patients may also undergo SPECT/CT at 15 and 28 days, and at 6 weeks based on whether there is uptake on prior imaging studies. Patients also undergo MRI, ultrasound imaging, blood sample collection and tissue biopsy throughout the trial.
  Interventions: Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter; Other: Quality-of-Life Assessment; Procedure: Single Photon Emission Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Ultrasound Imaging; Procedure: Biospecimen Collection; Procedure: Biopsy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Oncolytic Measles Virus Encoding Thyroidal Sodium Iodide Symporter — Given intratumorally
  Other Names: MV-NIS
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT imaging
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; Nuclear Magnetic Resonance Imaging; NMRI; Structural MRI; sMRI
Procedure: Ultrasound Imaging — Undergo ultrasound imaging
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: Bx
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and the best dose of a vaccine therapy in treating patients with malignant peripheral nerve sheath tumor that cannot be removed by surgery (unresectable) or has come back after a period of improvement (recurrent). Vaccines made from a gene-modified virus may kill tumor cells expressing a gene called neurofibromin 1 (NF1) without affecting surrounding normal cells and may also help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of intratumoral administration of an Edmonston strain measles virus genetically engineered to express neurofibromatosis type 1 (NIS) (oncolytic measles virus encoding thyroidal sodium iodide symporter [MV-NIS]) in patients with inoperable or recurrent malignant peripheral nerve sheath tumor (MPNST).

II. To determine the safety and toxicity of intratumoral administration of MV-NIS in patients with inoperable recurrent MPNST.

III. To preliminarily assess antitumor efficacy of intratumoral MV-NIS administration by the rate of progression-free survival at 3 months, achieved by following radiographic response of the treated lesion using World Health Organization (WHO) response criteria guidelines.

SECONDARY OBJECTIVES:

I. To determine the time course of viral gene expression and virus elimination and biodistribution of virally infected cells at various time points after infection with MV-NIS using single-photon emission computed tomography (SPECT)/computed tomography (CT) imaging.

II. To assess viremia, viral replication, and measles virus shedding/persistence following intratumoral administration.

III. To determine humoral and cellular immune response to the injected virus. IV. To assess the quality-of-life of patients treated with MV-NIS, using two inventories (Pain and Fatigue).

V. To assess time to progression and differences in growth rates between treated and untreated tumor lesions.

VI. To assess the overall survival time of patients treated with MV-NIS.

OUTLINE:

Patients receive MV-NIS intratumorally on day 1. Patients also undergo SPECT/CT at baseline and at 3 and 8 days after MV-NIS. Patients may also undergo SPECT/CT at 15 and 28 days, and at 6 weeks based on whether there is uptake on prior imaging studies. Patients also undergo magnetic resonance imaging (MRI), ultrasound imaging, blood sample collection and tissue biopsy throughout the trial.

After completion of study treatment, patients are followed up at 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Pathologically confirmed MPNST, with or without underlying diagnosis of neurofibromatosis type 1 (diagnostic criteria for neurofibromatosis type 1)
* Measurable disease as defined by at least one tumor that is measurable in two dimensions on CT or magnetic resonance imaging (MRI) scan (minimum size 1.0 cm for at least one lesion)
* MPNST for which standard therapy is not curative, including patients with surgically unresectable lesions, progression (WHO criteria) or recurrence of an MPNST in a previously radiated field (if it has been at least 4 weeks prior to registration since the last dose of radiation); Note: patients with metastatic disease also are eligible for participation
* Patient may have more than one site of recurrent or metastatic disease but only one lesion that is >= 1 cm in size will be injected (if in the lung, the lesion must be >= 2 cm and adjacent to the pleura in the lung)
* The following laboratory values obtained =< 14 days prior to registration

  * Absolute neutrophil count (ANC) >= 1500
  * Platelet (PLT) >= 100,000
  * Hemoglobin (HgB) >= 9.0 g/dL
  * Total bilirubin =< institutional upper limit of normal (ULN)
  * Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 1.5 x upper limit of normal (ULN)
  * Creatinine =< 1.0 mg/dL
  * International normalized ratio (INR) =< 2.0
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Provide informed written consent
* Willingness to return to Mayo Clinic Rochester for follow-up
* Willingness to provide biologic samples for correlative research purposes
* Life expectancy >= 12 weeks
* Cluster of differentiation (CD)4 count >= 200/uL or >= 15% of peripheral blood lymphocytes
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception during treatment and 8 weeks following the completion of treatment
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Receiving therapeutic anticoagulation (Coumadin or low molecular weight heparin, heparin, apixaban, dabigatran, rivaroxaban, warfarin)
* Active infection =< 5 days prior to registration
* History of tuberculosis or history of purified protein derivative (PPD) positivity
* Any of the following prior therapies:

  * Chemotherapy =< 3 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Biologic therapy =< 4 weeks prior to registration
  * Radiation therapy =< 3 weeks prior to registration
* Failure to fully recover from acute, reversible effects defined as =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.0 of prior chemotherapy regardless of interval since last treatment except alopecia and neuropathy
* Requiring blood product support
* Patient has central nervous system (CNS) metastases or seizure disorder. Note: Patients with seizures controlled by medication are eligible.
* Human immunodeficiency virus (HIV)-positive test result or history of other immunodeficiency
* History of organ transplantation
* History of chronic hepatitis B or C
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
* Treatment with oral/systemic corticosteroids, with the exception of topical or inhaled steroids
* Current exposure to household contacts =< 15 months old or household contact with known immunodeficiency; NOTE: patient must avoid contact during documented viral shedding; participants with continuous viral shedding will be given recommendations for restricted activities to avoid contact with immunocompromised persons
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination
* Allergy to iodine; Note: this does not include reactions to intravenous contrast materials
* Allergy to lidocaine, fentanyl, midazolam, or propofol (may be used during tumor biopsy or injection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Best response using the World Health Organization response criteria | From the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started), assessed up to 2 years
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and dose level).
Incidence of adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years after treatment
  The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Maximum tolerated dose defined as the highest safely tolerated dose level where at most 1 out of 6 patients experience dose-limiting toxicity (DLT) with the next higher dose having at least 2 patients out of a maximum of 6 patients experience DLT | 6 weeks
  Assessed according to according to Common Terminology Criteria for Adverse Events version 4.0. The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population.

SECONDARY OUTCOMES:
Absolute percentage change in quality of life measured using the Brief Pain Inventory (short form) and Brief Fatigue Inventory | Baseline to up to 2 years
  Determination of significant changes in quality of life over time will be assessed using a signed rank test comparing the change at each assessment point from baseline. Quality of life will be used as a descriptive supplement to other clinical information. Simple exploratory analysis may be undertaken to look for changes in quality of life scores over time as well as associations between change in quality of life scores at different time points and per dose level.
Change in biodistribution of virally infected cells at various time points after infection with MV-NIS using single photon emission computed tomography/computed tomography | Baseline to up to day 8
  Patients may be imaged on days 15, 28 and week 6. Absolute and percent change from baseline along with t-tests to evaluate change from baseline to all observed timepoints.
Growth-rate between treated and untreated lesions | Up to 2 years
  Differences in growth-rate between treated and untreated lesions will be compared using paired t-tests.
Humoral and cellular immune response to the injected virus | Up to 2 years
  Correlations between these laboratory values and other outcome measures will be carried out by standard parametric and nonparametric correlation procedures (Pearson's and Spearman's coefficients).
Incidence of measles virus shedding/persistence following intratumoral administration | Up to 2 years
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures like response, and dose levels will be carried out in an exploratory manner.
Incidence of viral replication following intratumoral administration | Up to 2 years
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures like response, and dose levels will be carried out in an exploratory manner.
Incidence of viremia following intratumoral administration | Up to 2 years
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures like response, and dose levels will be carried out in an exploratory manner.
Progression-free survival by radiographic response of the treated lesion using World Health Organization response criteria guidelines | At 3 months
  A progression-free survival at 3 months success is defined as a patient who is alive and their treated lesion is progression free at three months after they have treatment with oncolytic measles virus encoding thyroidal sodium iodide symporter (MV-NIS).
Time to progression | Up to 2 years
Time until hematologic nadirs (absolute neutrophil count, platelets, hemoglobin) | Up to 2 years
Viral gene expression | Up to 2 years
  Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Correlations between these laboratory values and other outcome measures like response, and dose levels will be carried out in an exploratory manner.
Virus elimination as monitored by single photon emission computed tomography/computed tomography imaging | Up to day 8
  Patients may be imaged on days 15, 28 and week 6. Descriptive statistics and simple scatterplots will form the basis of presentation of these data. Absolute and percent change from baseline along with t-Tests to evaluate change from baseline to all observed timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Dusica Babovic-Vuksanovic, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassan A, Pestana RC, Parkes A. Systemic Options for Malignant Peripheral Nerve Sheath Tumors. Curr Treat Options Oncol. 2021 Feb 27;22(4):33. doi: 10.1007/s11864-021-00830-7. PMID 33641042
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials